CLINICAL TRIAL: NCT04897360
Title: Effects of Hypocapnia on Postural Standing Balance Measured by Sharpened Romberg Testing (SRT) in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Sharpened Romberg Testing (SRT) in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jan Stepanek, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-012481
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hypocapnia; Balance; Distorted
Keywords: hypocapnia; balance
MeSH Terms: conditions — Hypocapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normocapnic SRT, Hypocapnic SRT, Recovery SRT (Experimental): Sharpened Romberg Test
  Interventions: Behavioral: Increased breathing; Other: sharpened Romberg test (SRT)

INTERVENTIONS:
Behavioral: Increased breathing — hyperventilation to lower ETCO2
Other: sharpened Romberg test (SRT) — Balance test conducted by standing with feet in front of each other, heel-to-toe in line while the right hand is on the left shoulder and the left hand is on the right shoulder.

SUMMARY:
This research study is being done to evaluate the effectiveness of using the sharpened Romberg test to screen for impaired postural control in patients with impaired or altered breathing patterns.

DETAILED DESCRIPTION:
The effects of hypocapnia on the postural system have not previously been adequately investigated. The specific aim of this study is to evaluate the effects of hypocapnia on postural standing balance using the sharpened Romberg test (SRT). There is very little research in this area, even though there is significant clinical relevance, ranging from individuals with conditions affecting ventilation (respiratory conditions, cardiac conditions, concussions, medications, post-surgical states requiring ventilatory support etc). The design of the experiment consists of testing healthy subjects and measuring their standing balance with SRT before and after they deliberately lower their carbon dioxide levels by increased ventilation over 2min. End-tidal CO2 (ETCO2) will be used to estimate the blood carbon dioxide level during the experimental procedures. ETCO2 will be measured using the Masimo, Emma Capnometer device. The device is a measurement tool that reads the end tidal carbon dioxide level on its display. The results will then be compared to the normal pre-hypocapnic SRT to assess how hypocapnia affects standing balance.

ELIGIBILITY:
Inclusion Criteria:

- Research subject conditions that may result in alterations of ventilatory control (capnic status) and balance will be specifically reviewed as criteria for participation.

Exclusion Criteria:

* Current pregnancy in women, alcohol use within the past 3 days prior to the experiment, history of balance problems (e.g., vertigo, neuropathy, central or peripheral vestibular disorders), and musculoskeletal disorders affecting the ability to perform a SRT in participants.
* Patients currently taking carbonic anhydrase inhibitors, opioids, benzodiazepines, hypnotics, first-generation H1 antihistamines, amphetamines, and first-generation antipsychotics.
* Patients with a history of insomnia, sleep apnea, circadian rhythm disturbances, narcolepsy, movement disorders, chronic low blood pressure, fainting spells, multiple concussions, seizure disorders, migraines, severe headaches and panic attacks.
* If the patient took medications known to cause prolonged QTc interval and other cardiac arrhythmias, the researchers will exclude the patient from the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Time to step out from sharpened Romberg test | approximately 10min
  measurement of time

SECONDARY OUTCOMES:
Capnic status | approximately 3 minutes
  measurement of ETCO2 with capnometer

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stepanek, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials